CLINICAL TRIAL: NCT02291042
Title: Pre-operative Administration of a Muscarinic Antagonist for Elective Cystoscopy Patients
Brief Title: Effect of an Anti-spasmodic Suppository to Improve Comfort After Urologic Surgery
Acronym: SPASMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern New Hampshire Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2014-05
Record Dates: First submitted 2014-10-13; First posted 2014-11-14 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Surgery
Keywords: Bladder; Surgery
MeSH Terms: interventions — Opium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Suppository (Experimental): Patients will receive a single antispasmodic muscarinic suppository after induction of anesthesia but before insertion of urological scope for surgery. The suppository is composed of Belladonna (16.2 mg) and Opium (30 mg) in a water soluble base manufactured as Belladonna and Opium Supprettes.
  Interventions: Drug: B+O Suppository
- Control (No Intervention): Patients will be provided with routine care.

INTERVENTIONS:
Drug: B+O Suppository
  Other Names: Belladona and opium; B+O Supprettes
  Arms: Suppository

SUMMARY:
This study evaluates the ability of a belladonna and opium suppository given prior to surgery to improve bladder comfort after surgery for patients who are having elective ureteroscopy surgery.

DETAILED DESCRIPTION:
Belladonna and opium suppositories are administered postoperatively to relieve bladder discomfort usually caused by bladder spasms. The onset of action of the suppository is 30-60 minutes. Bladder spasms are more likely to occur following uteroscopy procedures. The spasms result in a felt desire to void, even when there is no urine in the bladder. The spasms can produce pain or a sense of severe urgency.

By administering a belladonna and opium suppository at the beginning of surgery, it is hoped that there will be a decrease in the incidence of bladder spasms, increased comfort and less need for additional medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients from one urology practice schedule for elective uteroscopy.

Exclusion Criteria:

* Patients with pre-operative indwelling catheter or urinary stent.
* Patients who report any allergy to belladonna or opium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Difference in mean bladder comfort (baseline at PACU admission to PACU discharge) between experimental and control groups | Length of postoperative stay from admission to PACU to discharge from PACU an expected average of 2 hours
  Bladder comfort is defined as bladder pain and bladder urgency. Bladder pain is measured on a 0-10 verbal analog scale with 0 = no pain and 10 = most pain possible. Bladder urgency is measured by a 0 - 4 scale with 0 = no desire to void, 1 = awarenes of need to void which can be delayed at least 30 minutes, 2 = moderate urgency than can be delayed for no more than 15 minutes, 3 = severe urgency that can be delayed for no more than 5 minutes, 4 = must void now. Pain and urgency are reported by the patient with or without questioning by the nurse.

SECONDARY OUTCOMES:
Duration of PACU length of stay | Time from admission to PACU to discharge from PACU an expected average of 2 hours
  The time in minutes of the PACU length of stay

OTHER OUTCOMES:
Requirements for rescue therapy for pain and urgency | From PACU admission to PACU discharge an expected average of 2 hours
  Additional interventions for rescue pharmacology administered postoperatively to relieve pain or urgency

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Fetzer, PHD RN, Principal Investigator — Southern New Hampshire Medical Center

REFERENCES:
- [Background] Lukasewycz S, Holman M, Kozlowski P, Porter CR, Odom E, Bernards C, Neil N, Corman JM. Does a perioperative belladonna and opium suppository improve postoperative pain following robotic assisted laparoscopic radical prostatectomy? Results of a single institution randomized study. Can J Urol. 2010 Oct;17(5):5377-82. PMID 20974030
- [Background] Scavonetto F, Lamborn DR, McCaffrey JM, Schroeder DR, Gettman MT, Sprung J, Weingarten TN. Prophylactic belladonna suppositories on anesthetic recovery after robotic assisted laparoscopic prostatectomy. Can J Urol. 2013 Jun;20(3):6799-804. PMID 23783051